CLINICAL TRIAL: NCT01734798
Title: Adjuvant Post-radical Cystectomy Treatment for Bladder Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed s. Zaghloul, Professor of Radiation Oncology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Bladder-02
Record Dates: First submitted 2012-11-19; First posted 2012-11-28 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-11

CONDITIONS: Locally Advanced Bladder Cancer
Keywords: locally advanced bladder cancer; Postoperative radiotherapy; Adjuvant chemotherapy; Radical Cystectomy
MeSH Terms: interventions — Radiation; Gemcitabine; Cisplatin; Radiotherapy; Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (Experimental): post-operative radiotherapy will be done in locally advanced bladder cancer patients (P3b, P4a, G3 and / or LN positive patients) after radical cystectomy Dose of Radiotherapy: 45 Gray Gy/30 fractions/3 weeks
  Interventions: Radiation: Radiation
- Arm 2 (Experimental): adjuvant chemotherapy (gemcitabine and cisplatin) in addition to post operative radiotherapy in locally advanced bladder cancer patients (P3b, P4a, G3 and / or LN positive patients) after radical cystectomy
  Interventions: Other: Radiotherapy and Drug
- Arm 3 (Experimental): Adjuvant chemotherapy alone in locally advanced bladder cancer patients (P3b, P4a, G3 and / or LN positive patients) after radical cystectomy
  Interventions: Drug: gemcitabine and cisplatin

INTERVENTIONS:
Radiation: Radiation
  Arms: Arm 1
Drug: gemcitabine and cisplatin
  Arms: Arm 3
Other: Radiotherapy and Drug
  Arms: Arm 2

SUMMARY:
Radical Cystectomy is still the standard treatment in muscle-invasive Bladder cancer. Local recurrence is still the major cause of failure together with distant metastasis. postoperative radiotherapy succeeded to decrease the local recurrence and hence improved the overall survival. Adjuvant chemotherapy has also improved the survival in different studies. This study is performed to test the efficacy and toxicity of adding the two modalities together compared to each modality alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients not more than 70 years old.
* Radical cystectomy performed within 42 days with no microscopic or macroscopic residual after surgery (negative surgical safety margins)
* Having one or more of the risk factors ( P3b,P4a,G3 and /or positive LN)
* ECOG Performance Scale (0-2).
* Adequate liver functions.
* Adequate renal function serum (creatinine < 1.5 mg).
* No evidence of distant metastasis or other malignancy.

Exclusion Criteria:

* patients who received radiotherapy or chemotherapy prior to radical cystectomy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2002-12; Primary Completion 2008-01 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Comparison of the disease-free survival and overall survival of post-operative radiotherapy , adjuvant chemotherapy and the combined modalities [radiotherapy and chemotherapy] after radical cystectomy | Five-year overall and disease-free survival.
  Regular follow up is performed every 2 months in the first 2 years postcystectomy and every 6 months thereafter. Periodical CT pelvis is performed every 6 months in the first 2 years and yearly thereafter. The other appropriate radiological studies are performed in response to patients' symptoms and signs. Treatment side effects (immediate and late) are reported in each follow up visit.

SECONDARY OUTCOMES:
comparison of the Local recurrence rate in the three Arms | Five year local pelvic control rate
  Periodical CT pelvis is performed every 6 months in the first 2 years and yearly thereafter. The other appropriate radiological studies are performed in response to patients' symptoms and signs. Treatment side effects (immediate and late) are reported in each follow up visit.

CONTACTS AND LOCATIONS:
Locations (1):
- National cancer Institute-Cairo University, Cairo, Egypt

REFERENCES:
- [Derived] Zaghloul MS, Christodouleas JP, Smith A, Abdallah A, William H, Khaled HM, Hwang WT, Baumann BC. Adjuvant Sandwich Chemotherapy Plus Radiotherapy vs Adjuvant Chemotherapy Alone for Locally Advanced Bladder Cancer After Radical Cystectomy: A Randomized Phase 2 Trial. JAMA Surg. 2018 Jan 17;153(1):e174591. doi: 10.1001/jamasurg.2017.4591. Epub 2018 Jan 17. PMID 29188298